CLINICAL TRIAL: NCT02644577
Title: Metformin for Treatment Antipsychotic-induced Metabolic Syndrome in Bipolar Disorder Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Man Wang, Associate Professor of department of psychiatry, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MWang-BD1
Record Dates: First submitted 2015-12-29; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Bipolar Disorder
Keywords: Metformin; antipsychotic-induced metabolic syndrome; bipolar disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Metformin; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metformin group (Experimental): Metformin 1000mg/day
  Interventions: Drug: Metformin
- placebo group (Placebo Comparator): starch
  Interventions: Other: Starch

INTERVENTIONS:
Drug: Metformin
  Arms: metformin group
Other: Starch
  Arms: placebo group

SUMMARY:
The purpose of this study is to test the efficacy of metformin for treatment antipsychotic-induced metabolic syndrome in bipolar disorder patients.

DETAILED DESCRIPTION:
Patients aged 18 to 45 years with bipolar disorder diagnosed in accordance with criteria set out in the Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV) were eligible for our study, and the Structured Clinical Interview of DSM-IV Axis I Disorders (SCID-1), Clinical Version, was used during the screening phase. To be qualified for this study, patients had to meet, 1) have experienced metabolic syndrome as defined below within the first year of treatment with one of four antipsychotics-clozapine, olanzapine, risperidone, or sulpiride; 2) had been either discharged from inpatient units or first visit in the outpatient clinic in the 12 months before enrollment, and their glucose and lipid levels, weight, blood pressure and antipsychotic treatment were documented; 3) had taken single antipsychotic medication, with no more than a 25% change in dosage, over the past 3 months. All participants had to be under the care of a parent or another adult caregiver who monitored and recorded the intake of medication daily during the trial to assure the adherence to medication. Patients were excluded from the study if there was evidence of liver or renal dysfunction, cardiovascular disease, or diabetes mellitus; or if they were pregnant or lactating; or had any psychiatric diagnosis other than schizophrenia.

The primary outcome was the level of LDL-C or the percentage of patients who had LDL-C greater or equal 3.37mmol/L (130mg/dl). The secondary outcomes were fasting triglyceride, total cholesterol, HDL-C, insulin and glucose levels, insulin resistance index, body weight and body mass index, as well as incidence of adverse events. Body mass index was calculated as weight in kilograms divided by height in meters squared. Insulin resistance index was calculated based on the homeostasis model assessment as: fasting insulin (mIU/L)×fasting glucose (mmol/L)/22.5. the assessment was conducted by members of a trained independent research team connected to the centre. Inclusion or exclusion was decided by the team. After a complete description of the study to the subjects, written informed consent was obtained in accordance with National Health and Medical Research Council guidelines.

ELIGIBILITY:
* Inclusion Criteria:

  * clinical diagnosis of bipolar disorder
  * have experienced metabolic syndrome as defined below within the first year of treatment with one of four antipsychotics-clozapine, olanzapine, risperidone, or sulpiride
  * had been either discharged from inpatient units or first visit in the outpatient clinic in the 12 months before enrollment, and their glucose and lipid levels, weight, blood pressure and antipsychotic treatment were documented
  * had taken single antipsychotic medication, with no more than a 25% change in dosage, over the past 3 months
  * must be under the care of a parent or another adult caregiver who monitored and recorded the intake of medication daily during the trial to assure the adherence to medication
* Exclusion Criteria:

  * any psychiatric diagnosis other than schizophrenia
  * liver dysfunction
  * renal dysfunction
  * cardiovascular disease
  * diabetes mellitus
  * pregnancy
  * lactation period

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2012-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
the percentage of patients who had metabolic syndrome | week 24

SECONDARY OUTCOMES:
body mass index | week 24
blood pressure | week 24
fasting glucose | week 24
lipid levels | week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, the First Hospital of China Medical University, Shenyang, Liaoning, China